CLINICAL TRIAL: NCT01830907
Title: Efficacy of Preoperative Nutritional Support on Postoperative Outcome in Gastric Cancer Patients at Nutritional Risk by NRS-2002- A Prospective, Randomized Clinical Trial
Brief Title: Efficacy of Preoperative Nutritional Support on Postoperative Outcome in Gastric Cancer Patients at Nutritional Risk by NRS-2002
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Punyaram Kharbuja, MD, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: First Hospital of JLU
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Malnutrition; Gastric Cancer
Keywords: Malnutrition; Gastric cancer; preoperative nutrition
MeSH Terms: conditions — Malnutrition; Stomach Neoplasms | interventions — Carbohydrates; Vitamins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enteral (Active Comparator): Enteral nutrition composed of carbohydrates and vitamins
  Interventions: Dietary Supplement: carbohydrates; Dietary Supplement: vitamins
- Parenteral (Active Comparator)
  Interventions: Dietary Supplement: carbohydrates; Dietary Supplement: vitamins

INTERVENTIONS:
Dietary Supplement: carbohydrates
Dietary Supplement: vitamins

SUMMARY:
Evaluation of the impact of preoperative nutritional support on clinical outcomes in patients at nutritional risk. The primary endpoint was the complication rate and the second endpoint was the length of stay.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of gastric cancer surgery preoperative stage

Exclusion Criteria:

* neoadjuvent chemoradiation
* pregnant
* advanced stage

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Infectious complication | 30 days

SECONDARY OUTCOMES:
Length of hospital stay | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- First hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Background] van Stijn MF, Korkic-Halilovic I, Bakker MS, van der Ploeg T, van Leeuwen PA, Houdijk AP. Preoperative nutrition status and postoperative outcome in elderly general surgery patients: a systematic review. JPEN J Parenter Enteral Nutr. 2013 Jan;37(1):37-43. doi: 10.1177/0148607112445900. Epub 2012 May 1. PMID 22549764